CLINICAL TRIAL: NCT01395888
Title: A 12 Week Study to Evaluate the Effect of Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) 100/25 mcg Inhalation Powder Delivered Once Daily Via a Novel Dry Powder Inhaler (NDPI) on Arterial Stiffness Compared With Tiotropium Bromide 18 mcg Delivered Once Daily Via a HandiHaler in Subjects With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Study to Compare the Impact of Fulticasone Furoate/Vilanterol vs. Tiotropium on Arterial Stiffness in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115247
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relovair (Experimental): Inhaled long-acting bronchodilator and corticosteroid combination
  Interventions: Drug: fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) 100/25 mcg Novel Dry Powder Inhaler (NDPI)
- Tiotropium (Active Comparator): Inhaled long-acting anticholinergic
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) 100/25 mcg Novel Dry Powder Inhaler (NDPI) — fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) 100/25 mcg Inhalation Powder delivered once daily via a Novel Dry Powder Inhaler (NDPI)
  Arms: Relovair
Drug: Tiotropium — • Tiotropium (18 mcg) administered QD via a HandiHaler
  Arms: Tiotropium

SUMMARY:
This study is designed to evaluate the effect of fluticasone furoate (FF, GW685698)/vilanterol (VI, GW642444) Inhalation Powder once daily (QD) on arterial stiffness compared with Tiotropium QD over 12 week treatment period in subjects with COPD and aortic pulse wave velocity (aPWV) > 12.0 m/s at Visit 1. Arterial stiffness will be measured as aPWV. This is a comparator, randomised, double-blind, double-dummy, parallel group, multi-centre study. Subjects who meet the eligibility criteria at Screening and meet the randomization criteria at the end of a 2-week Run-In period will enter a 12-week treatment period. There will be an approximate 7-day Follow-up period after the treatment period.

DETAILED DESCRIPTION:
This is a Phase IIIb comparator, double-blind, double-dummy, randomised (1:1), parallel group, multi-centre study. At Visit 1 (Screening Visit), subjects who meet the pre-defined Inclusion Criteria and none of the Exclusion Criteria will enter a 2-week, single-blind placebo Run-in Period. The purpose of the Run-In Period is to monitor albuterol/salbutamol use at baseline, and to ensure that subjects' COPD is at a stable stage at randomization. Subject's adherence with study procedures, diary completion will also be evaluated during the Run-In Period. At the end of the Run-in period, subjects will be assessed and those who meet the randomisation criteria will receive one of the following two double-blind treatments for 12 weeks:

* FF (100 mcg)/VI (25 mcg) administered QD via a NDPI in the morning
* Tiotropium (18 mcg) administered QD via a HandiHaler in the morning

To ensure blinding of the treatments and to ensure a double-dummy design matching NDPI and HandiHaler will be utilised. Each subject will be instructed to self administer blinded study drug during the double blind treatment period as follows:

* Each morning take 1 inhalation from NDPI containing FF (100 mcg)/VI (25 mcg) followed by 1 inhalation from placebo capsule delivered via HandiHaler.
* Each morning take 1 inhalation from matching placebo NDPI followed by 1 inhalation from a capsule containing tiotropium 18 mcg delivered via HandiHaler.

An inhaled short acting beta2-receptor agonist, salbutamol/albuterol will be provided to subjects to use as needed throughout the Run-in and Treatment periods for relief of COPD symptoms. Ipratropium bromide is permitted if the subject is on a stable dose from Screening (Visit 1) and remains on the stable dose throughout the study. Subjects who experience an exacerbation of their COPD (which requires medication in addition to an increase in rescue medication) or a lower respiratory tract infection (LRTI) during the run-in period are not eligible to enter the treatment period. Any subject who experiences a similar COPD exacerbation (sec 4.4) or LRTI at any time on therapy will be withdrawn from the study. The aPWV will be measured at Screening and clinic Visits 3-5. Disease specific health status will be evaluated using the St. George's Respiratory Questionnaire (SGRQ-C), Euro Qol Questionnaire (EQ-5D) for COPD patients and the COPD Assessment Test (CAT) at Visit 2 (Day 1) and at Visit 5 (Weeks 12). The 12-lead ECG will be evaluated at Visit 1 (Screening) only. Vital signs (blood pressure and pulse rate), spirometry measurements, and clinical laboratory tests (hematology and chemistry) and other study-specific safety assessments will be obtained at selected clinic visits. A follow-up phone call will occur approximately 7 days after the last clinic visit. The overall study duration from Screening to Follow-up for each subject is approximately 15 weeks. Subjects will be considered to have completed the study upon completion of assessments and procedures up to and including completion of Follow-up Phone Contact (7 ± 2 days post Visit 5).

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Male or female subjects.
* Age: greater then or equal to 40 years of age at Screening (Visit 1)
* COPD diagnosis: Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society (ATS) /European Respiratory Society(ERS).
* Subjects with a current or prior history ofgreater then or equal to 10 pack-years of cigarette smoking at Screening (Visit 1).
* Subjects with a measured post-albuterol/salbutamol FEV1 less then 70% of predicted at Screening (Visit 1).
* Subjects with a measured post-albuterol/salbutamol FEV1/FVC ratio of less then or equal to 0.70 at Screening (Visit 1).
* Exacerbation History: Subjects who have been hospitalised or have been treated with oral corticosteroids or antibiotics for their COPD within the last 3 years prior to Screening (V1).
* Baseline aPWV: subjects with a measured aPWV greater then 12.0 m/s at Screening (Visit 1).

Exclusion Criteria:

* Body Mass Index of less then or equal to 35

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-06-30; Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (45):
- Argentina (6):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, San Miguel de Tucumán
- France (6):
  - GSK Investigational Site, Béthune
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Saint-Michel
- Germany (8):
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (5):
  - GSK Investigational Site, Cassano Murge (BA), Apulia
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Crema, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
- Norway (4):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Skedsmokorset
- Russia (10):
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kokhma
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Vladivostok, Primorskiy Kray
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- Ukraine (6):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Yalta

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pepin JL, Cockcroft JR, Midwinter D, Sharma S, Rubin DB, Andreas S. Long-acting bronchodilators and arterial stiffness in patients with COPD: a comparison of fluticasone furoate/vilanterol with tiotropium. Chest. 2014 Dec;146(6):1521-1530. doi: 10.1378/chest.13-2859. PMID 25058845
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 260 participants were randomized. Three of these participants were randomized in error (they were determined not to have met entry criteria and were classified as run-in/screen failures); thus, they did not receive investigational product and are not captured in the Treatment Period table of the Participant Flow module.
Pre-assignment Details: At Visit (V) 1, eligible participants (par.) entered a 2-week, single-blind placebo Run-in Period (RIP) to establish a stable baseline. At V 2, eligible par. were randomized to a 12-week, double-blind, double-dummy Treatment Period. 802 par. were screened, 279 par. entered the RIP, and 257 par. were randomized and received >=1 study treatment dose.
Groups:
- Salb/Alb + IBr: Participants were provided with an inhaled short-acting beta2-receptor agonist, salbutamol/albuterol (Salb/Alb), for use as needed throughout the Run-in Period for relief of chronic obstructive pulmonary disease (COPD) symptoms. Ipratropium bromide (IBr) was permitted during the Run-in Period and for up to 4 hours prior to Randomization (Visit 2) if the participant was on a stable dose prior to Screening (Visit 1). Following randomization, IBr was not permitted during exposure to study treatment.
- FF/VI 100/25 µg: Participants (par.) self-administered one inhalation of Fluticasone Furoate /Vilanterol (FF/VI) 100/25 micrograms (µg) via a dry powder inhaler (DPI) followed by 2 inhalations from a single placebo capsule delivered via a HandiHaler in the morning for 12 weeks. An inhaled short-acting beta2-receptor agonist, salbutamol/albuterol, was provided for participants to use as needed throughout the Treatment Period for relief of Chronic Obstructive Pulmonary Disease (COPD) symptoms.
- Tiotropium Bromide 18 µg: Participants self-administered one inhalation of placebo via an DPI followed by 2 inhalations from a single capsule containing Tiotropiuum Bromide 18 µg via a HandiHaler. An inhaled short-acting beta2-receptor agonist, salbutamol/albuterol, was provided for participants to use as needed throughout the Treatment Period for relief of COPD symptoms.
Period: 2-week Run-in Period
Arm/Group | Salb/Alb + IBr | FF/VI 100/25 µg | Tiotropium Bromide 18 µg
Started | 279 | 0 | 0
Completed | 257 | 0 | 0
Not Completed | 22 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Continuation Criteria Not Met | 13 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Treatment Period (TP)
Arm/Group | Salb/Alb + IBr | FF/VI 100/25 µg | Tiotropium Bromide 18 µg
Started | 0 | 127 | 130
Completed the Treatment Period | 0 | 112 (Participants were considered to have completed the TP if they attended Visit 5 (Week 12).) | 113 (Participants were considered to have completed the TP if they attended Visit 5 (Week 12).)
Completed | 0 | 112 (Par. completed the study if they completed the TP and a safety follow-up phone contact 1 week later.) | 113 (Par. completed the study if they completed the TP and a safety follow-up phone contact 1 week later.)
Not Completed | 0 | 15 | 17
Not completed — Adverse Event | 0 | 7 | 6
Not completed — Lack of Efficacy | 0 | 4 | 3
Not completed — Protocol Violation | 0 | 1 | 5
Not completed — Met Protocol-defined Stopping Criteria | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- FF/VI 100/25 µg: Participants self-administered one inhalation of Fluticasone Furoate /Vilanterol (FF/VI) 100/25 micrograms (µg) via a dry powder inhaler (DPI) followed by 2 inhalations from a single placebo capsule delivered via a HandiHaler in the morning for 12 weeks. An inhaled short-acting beta2-receptor agonist, salbutamol/albuterol, was provided for participants to use as needed throughout the Treatment Period for relief of Chronic Obstructive Pulmonary Disease (COPD) symptoms.
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg | Tiotropium Bromide 18 µg | Total
Number analyzed (Participants) | 127 | 130 | 257
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (7.20) | 67.7 (7.34) | 67.3 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 108 | 112 | 220
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European | 127 | 130 | 257

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) in Aortic Pulse Wave Velocity (aPWV) at the End of the 12-week Treatment Period (Day 84)
Description: PWV is defined as the speed of travel of the pressure pulse along an arterial segment and can be obtained for any arterial segment accessible to palpation. aPWV is measured with tonometers positioned transcutaneously at the base of the common carotid artery and over the femoral artery. PWV increases with arterial stiffness and is defined by the Moens-Korteweg equation: PWV=square root of Eh/2pR, where E is Young's modulus of the arterial wall, h is the wall thickness, R is the arterial radius at the end of diastole, and p is the blood density. Change from Baseline was calculated as the Day 84 value minus the Baseline value. The analysis was performed using a repeated measures model with covariates of treatment, visit, age, gender, smoking status at screening, geographical region, Baseline aPWV, and interaction terms of Baseline by visit and treatment by visit.
Time Frame: Baseline to Day 84 (Early Withdrawal)
Population: Intent-to-Treat (ITT) Population: all participants (par.) who were randomized to and received >=1 dose of randomized medication in the TP. The analysis model included all par. in the ITT Population without missing covariate information (MCI) and with >=1 post-BL measurement. Par. presented represent those with data available at Day 84 without MCI.
Measure: Least Squares Mean (Standard Error); unit: meters per second (m/sec)
Arm/Group | FF/VI 100/25 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 106 | 102
meters per second (m/sec) | -0.859 (0.2590) | -1.118 (0.2620)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.484, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.259, 95% CI 2-sided [-0.468 to 0.986]

ADVERSE EVENTS:
Arm/Group | FF/VI 100/25 µg | Tiotropium Bromide 18 µg
Serious Adverse Events (participants affected / at risk) | 7/127 | 8/130
Other Adverse Events (participants affected / at risk) | 8/127 | 8/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg (N=127) | Tiotropium Bromide 18 µg (N=130)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg (N=127) | Tiotropium Bromide 18 µg (N=130)
Nasopharyngitis (Infections and infestations) | 5 | 4
Headache (Nervous system disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.